CLINICAL TRIAL: NCT00271713
Title: Randomized Double-Blind Placebo-Controlled and Parallel Group Study to Evaluate the Impact of One Year Therapy With Monthly Oral Ibandronate 150 mg on Structural Properties of Bone in Postmenopausal Osteoporosis Without Vertebral Fractures
Brief Title: Impact of Oral Ibandronate 150 mg Monthly on Structural Properties of Bone in Postmenopausal Osteoporosis (SPIMOS-3D)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Charite University, Berlin, Germany, center for muscle and bone research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ML 19472
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: bone structure; ibandronate
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibandronate (Active Comparator): 150 mg ibandronate monthly plus 500mg calcium and 800 UI vitamin D daily
  Interventions: Drug: ibandronate, calcium and vitamin D
- 2 (Placebo Comparator): placebo monthly plus 500mg calcium and 800 UI vitamin D daily
  Interventions: Drug: placebo,calcium and vitamin D

INTERVENTIONS:
Drug: ibandronate, calcium and vitamin D — 1: 150 mg ibandronate monthly plus 500mg calcium and 800 UI vitamin D daily or
  Arms: ibandronate
Drug: placebo,calcium and vitamin D — 2: placebo monthly plus 500mg calcium and 800 UI vitamin D daily
  Arms: 2

SUMMARY:
Efficacy:

To investigate changes of structural bone properties in vivo using 3DpQCT ("Xtreme" CT, Scanco) in monthly oral ibandronate therapy for women with postmenopausal osteoporosis.

Major structural bone parameters which determine bone strength and predict fracture risk earlier and more precisely are measurable in vivo by 3DpQCT.

Safety:

To assess the tolerability and safety of ibandronate therapy

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 75 years
* Menopause > 5 years
* Spine (L1 - L4) or hip BMD ≤ -2.0 and > -3.5 SD T-score measured by DXA
* Patients who, in the opinion of the investigator, are able and willing to comply with the protocol for its duration
* Written informed consent
* 3DpQCT measurable at both skeletal sites, distal tibia and radius

Exclusion Criteria:

* Spine or hip BMD ≤ -3,5 SD T-Score measured by DXA
* Vertebral fractures
* Multiple (>2) low trauma peripheral fractures
* Disease/disorder known to influence bone metabolism
* History of major upper gastro-intestinal (GI) disease
* Diagnosed malignant disease within the previous 10 years
* Previous treatment with a bisphoshonate at any time
* Treatment with fluoride for osteoporosis (dose greater than 10 mg/day) within the last 12 months, or for more than 2 years (total duration)
* Treatment with PTH and similar agents or strontium ranelate at any time
* Treatment with other drugs affecting bone metabolism within the last 6 months
* Chronic systemic corticosteroid treatment
* Estrogens, progestins, SERMs, anabolic steroids, active vitamin D analogues/metabolites, calcitonin
* Calcineurin inhibitors (e.g. cyclosporine, tacrolimus) or methotrexate
* Total serum calcium < 2.2 mmol/l or > 2.6 mmol/l
* Vitamin D deficiency (serum 25-hydroxy vitamin D < 12 ng/ ml)
* ALT above triple upper limit of normal range
* Renal impairment (serum creatinine > 210 µmol/l)
* Contra-indications for ibandronate, calcium or vitamin D
* Employees of the Centre for Muscle and Bone Research, or their relatives

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
BV/TV and trab. Sp. measured by 3D pQCT device | Baseline and after 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Felsenberg, Prof. Dr., Principal Investigator — Centre for Muscle and Bone Research, Charité - Campus Benjamin Franklin, Berlin, 12200, Germany
Locations (1):
- Centre for Muscle and Bone Research, Charité - Campus Benjamin Franklin, Berlin, Germany